CLINICAL TRIAL: NCT01964911
Title: Monocentric Prospective Study, in Order to Assess Analgesia Provided by Continuous Sciatic Nerve Block, in Patients With Hypertensive Leg Ulcer.
Brief Title: To Assess Analgesia Provided by Continuous Sciatic Nerve Block in Patients With Hypertensive Leg Ulcer
Acronym: ANGIOCATH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC13_0252
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Hypertensive Leg Ulcer
Keywords: Martorell ulcer; Hypertensive leg ulcer; Pain; Continuous nerve block; Ropivacaïne; Local anesthesic
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ropivacaïne (Experimental)
  Interventions: Drug: Ropivacaïne

INTERVENTIONS:
Drug: Ropivacaïne — The first 3 days, analgesic treatments will be provided, as usual, depending on pain intensity (EN <3/10 : non opioids, EN 3-5/10 : weak opioids, EN>5/10 : strong opioids).
  If NRS is still over 5/10, continuous nerve block will be proposed. Patients will receive ropivacaïne, 5 mL/h during 7 days, with possibility of one bolus before wound care, through a stimulating catheter stimulong sono®.
  In association, analgesic treatments will be provided, as usual, depending on pain intensity (as during the first 3 days).

SUMMARY:
Hypertensive leg ulcer, also called Martorell ulcer, represents 1 to 15% of leg ulcers in hospital. These ulcers are painful, long to heal, and hospitalization is sometimes necessary for analgesia and debridement of necrotic tissue. Strong opioids are often required, and are responsible of many side effects. Martorell ulcer arises predominantly in women over 60 years of age, with history of vascular disease, and therefore with a higher risk of adverse event. Pain is also part of the physiopathology, inducing a vasospasm which increases ulcer extension and ischemia.

This is why pain management is one of the main challenge in treatments of these ulcers.

Continuous nerve block of lower limbs are often used during per and postoperative orthopaedic surgery. Few adverse events and rare serious adverse events related to local anesthesic are reported (respectively <1% and <1/1000), and few adverse events related to catheter are reported (<1%). Its benefits have been proved on post-operative pain management and reeducation.

The aim of this study is to assess analgesia provided by continuous sciatic nerve block, in patients with hypertensive leg ulcer, during hospitalization.

Thirty patients will be enrolled on a 3-years period. They will receive a continuous sciatic nerve block with ropivacaïne 0,2%, during 7 days.

Pain intensity will be assessed by 4 datas : numerating rating scale (NRS) at rest, during wound care, maximal and mean. These datas will be collected over two 3-days period : the first 3 days of hospitalization, in which pain treatment will be prescribed depending on pain intensity of the patient ; and the first 3 days of ropivacaïne treatment.

The main evaluation criteria will be at least a 50% decrease of one of the pain NRS when receiving ropivacaïne.

Time to healing, microcirculation evolution measured by Transcutaneous Oxygen Pressure (TcPO2), and quality of life of patients will be collected over a 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Hospitalized for hypertensive leg ulcer with severe pain :
* For which pain intensity has been collected over the first 3 days before catheter insertion (D0)
* With severe pain (mean or at wound care) in spite of acetaminophen treatment (NRS ≥ 5/10), and/or with adverse events related to weak or strong opioids.
* patients' written informed consent obtained

Exclusion Criteria:

* Patients with moderate pain after 3 days of usual pain management in hospitalization : mean NRS<5/10 the 24 hours before D0
* pregnant women
* other ulcer causes, local or systemic infection
* not able to provide informed consent or to answer the pain evaluation
* dialysis patients
* unstable active diseases
* Charcot foot
* Known allergy to any local anesthetics
* Ankle-brachial index <0,6
* hemodynamically significant stenosis on arterial Doppler ultrasound
* current clopidogrel or prazugrel treatment the 10 days preceding catheter insertion
* current clopidogrel or prazugrel treatment the 10 days preceding catheter insertion, with contraindication to salicylic acid
* current anticoagulant treatment, with contraindication to LMWHs or UFH

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
number of patient with a 50% decrease of one of the pain NRS | 3 days
  The main evaluation criteria will be at least a 50% decrease of one of the pain NRS (at rest, during wound care, maximal or mean) with 3 days of ropivacaïne treatment, compared to 3 days of usual analgesic treatment.

SECONDARY OUTCOMES:
Evolution of NRS | 6 month
  NRS during the 7 days of ropivacaïne, and during the 6 months follow up
To assess patients's satisfaction with Patient Global Impression of Change | 6 month
To assess quality of life using Short Form 36 (SF36) | 6 month
  Quality of life using a standardized questionnaire : SF36
To assess pain consequences using Hospital Anxiety and Depression Scale (HAD) and Brief Pain Inventory questionnaire(BPI) | 6 month
  Pain consequences using standardized questionnaire : HAD, BPI
To assess microcirculatory evolution with a TCPO2 measure | 6 month
  Microcirculatory evolution with a TCPO2 measure before and after ropivacaïne treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cécile DURANT, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France